CLINICAL TRIAL: NCT04323098
Title: A Phase 3b, Single Arm, Open-Label Study to Evaluate the Efficacy and Safety of BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII, With Prophylactic Corticosteroids in Hemophilia A Patients
Brief Title: Study to Evaluate the Efficacy and Safety of Valoctocogene Roxaparvovec, With Prophylactic Steroids in Hemophilia A
Acronym: GENEr8-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-303
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
Keywords: Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases; Factor VIII; Coagulants
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- valoctocogene roxaparvovec (Experimental): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg with prophylactic corticosteroids
  Interventions: Biological: valoctocogene roxaparvovec

INTERVENTIONS:
Biological: valoctocogene roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
  Other Names: BMN 270

SUMMARY:
This Phase III clinical study will evaluate the safety and effectiveness of valoctocogene roxaparvovec in combination with prophylactic corticosteroids in patients with severe hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Males >= 18 years of age with hemophilia A and residual FVIII levels <= 1 IU/dL as evidenced by medical history, at the time of signing the informed consent.
2. Must have been on prophylactic hemophilia therapy for at least 12 months prior to study entry. High-quality, well-documented historical data concerning bleeding episodes and hemophilia therapy usage over the previous 12 months must be available.
3. Treated/exposed to FVIII concentrates or cryoprecipitate for a minimum of 150 exposure days (EDs).
4. Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any study-related procedures.
5. No previous documented history of a detectable FVIII inhibitor, and results from a Bethesda assay or Bethesda assay with Nijmegen modification of less than 0.6 Bethesda Units (BU) (or less than 1.0 BU for laboratories with a historical lower sensitivity cutoff for inhibitor detection of 1.0 BU) on 2 consecutive occasions at least one week apart within the past 12 months (at least one of which should be tested at the central laboratory).
6. Sexually active participants must agree to use an acceptable method of effective contraception, either double-barrier contraception (ie, condom + diaphragm; or condom or diaphragm + spermicidal gel or foam) or their female partner either using hormonal contraceptives or having an intrauterine device. Participants must agree to contraception use for at least 12 weeks post-infusion; after 12 weeks, participants may stop contraception use only if they have had 3 consecutive semen samples with viral vector DNA below the limit of detection.
7. Willing to abstain from alcohol consumption for at least the first 52 weeks following BMN 270 infusion.

Exclusion Criteria:

1. Participants with detectable pre-existing antibodies to the adeno-associated virus (AAV5) capsid are excluded with the following exception: up to 25% of participants may have detectable pre-existing AAV5 capsid antibodies with titer level below the minimum required dilution (< 20).
2. Any evidence of active infection, including Coronavirus Disease (COVID-19), or any immunosuppressive disorder, except for HIV infection. HIV-positive patients who meet all other eligibility criteria may be included if they have a CD4 count > 200/mm^3 and an undetectable viral load (unquantifiable viral load as defined as less than the limit of quantification by the testing laboratory's assay is permitted) while receiving an antiretroviral therapy (ART) regimen that does not contain efavirenz or another potentially hepatotoxic ART.
3. Significant liver dysfunction with any of the following abnormal laboratory results: alanine aminotransferase (ALT) > 1.25x upper limit of normal (ULN);aspartate aminotransferase (AST) > 1.25x ULN;gamma-glutamyltransferase (GGT) > 1.25x ULN;Total bilirubin > 1.25x ULN;Alkaline phosphatase > 1.25x ULN; or international normalized ratio (INR) >= 1.4.

   Participants whose liver laboratory assessments fall outside of these ranges could undergo repeat testing of the entire liver test panel within the same Screening window and, if eligibility criteria are met on retest, could be enrolled after confirmation by the Medical Monitor.
4. FibroScan or prior liver biopsy showing significant fibrosis of 3 or 4 as rated on a scale of 0-4 on the Batts-Ludwig (Batts 1995) or METAVIR (Bedossa 1996) scoring systems, or an equivalent grade of fibrosis if an alternative scale is used.
5. Evidence of any bleeding disorder not related to hemophilia A.
6. Platelet count of < 100 x 10^9/L.
7. Creatinine >= 1.5 mg/dL
8. Liver cirrhosis or other clinically significant liver disease of any etiology as assessed by FibroScan or liver ultrasound.
9. Chronic or active hepatitis B as evidenced by positive serology testing (hepatitis B surface antigen [HBsAg], hepatitis B surface antibody [HBsAb], and hepatitis B core antibody [HBcAb]) and confirmatory hepatitis B virus (HBV) DNA testing. Refer to the Centers for Disease Control (CDC) table for the interpretation of serological test results in the Laboratory Manual.
10. Active Hepatitis C as evidenced by detectable hepatitis C virus (HCV) RNA or currently on antiviral therapy.
11. Active malignancy, except non-melanoma skin cancer.
12. History of hepatic malignancy.
13. History of arterial or venous thromboembolic events (eg, deep vein thrombosis, non-hemorrhagic stroke, pulmonary embolism, myocardial infarction, arterial embolus), with the exception of catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing.
14. Known inherited or acquired thrombophilia, including conditions associated with increased thromboembolic risk, such as atrial fibrillation.
15. Treatment with any investigational product within 30 days or 5 half-lives of the investigational product prior to the screening period. For participants who have received a prior investigational product, all ongoing adverse events (AEs) experienced while receiving that investigational product must have resolved prior to screening for this study.
16. Any condition that, in the opinion of the Investigator or Sponsor would prevent the patient from fully complying with the requirements of the study (including possible corticosteroids (CS) treatment and/or use of alternative immunosuppressive agents (AIS) outlined in the protocol) and/or would impact or interfere with evaluation and interpretation of participant safety or efficacy result.
17. Prior treatment with any vector or gene transfer agent.
18. Major surgery planned in the 52-week period following the infusion with BMN 270.
19. Use of systemic immunosuppressive agents, not including CS, or live vaccines within 30 days before the BMN 270 infusion.
20. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study that does not interfere with the requirements of the current protocol or have the potential to impact the evaluation of efficacy and safety of BMN 270 and with prior consultation with the Medical Monitor.
21. Known allergy or hypersensitivity to BMN 270 investigational product formulation.
22. Unwilling to receive blood or blood products for treatment of an adverse event and/or a bleeding episode.

Optional Liver Biopsy Inclusion and Exclusion Criteria

Individuals eligible for the optional liver biopsy must meet the following inclusion criteria:

1. Able to sign informed consent and comply with requirements for the optional liver biopsy
2. Documentation of FVIII activity >= 50 IU/dL (or higher, depending on local guidelines and/or Investigator discretion) within 24 hours prior to the liver biopsy being performed (FVIII activity levels should be assessed at the local laboratory). Participants may be treated with additional exogenous FVIII replacement products in order to increase their FVIII activity to an appropriate level, under the supervision/instruction of the Investigator.

Individuals who meet the following exclusion criterion are not be eligible for the optional liver biopsy:

1. Any condition that, in the opinion of the Investigator or a hepatologist/radiologist would make liver biopsy contraindicated. This includes (but is not limited to) abnormalities detected on liver ultrasound performed within 28 days of procedure, or prior liver ultrasound result within 90 days that would preclude safe performance of the biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males only
Enrollment: 22 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (12):
- United States (3):
  - University of California Davis Health, Sacramento, California
  - Washington University School of Medicine, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
- Australia (5):
  - The Royal Adelaide Hospital, Adelaide
  - Royal Brisbane and Women's Hospital, Brisbane
  - Alfred Hospital, Melbourne
  - Fiona Stanley Hospital, Perth
  - Royal Prince Alfred Hospital, Sydney
- Brazil (2):
  - Campinas University Clinical Hospital, Campinas
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Taiwan (2):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Taichung Veterans General Hospital, Taichung

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by 12 principal investigators at 12 study centers in 4 countries (United States, Australia, Brazil, and Taiwan)
Pre-assignment Details: Total of 34 subjects were screened. Of these, 12 subjects failed screening and remaining 22 subject was enrolled in the study. Of the 22 enrolled participants, all 22 completed the Week 52 visit, and all 22 remained enrolled in the study as on data cut-off date 27January2023.
  While up to 25% of patients could be AAV5+, no such patients were enrolled, i.e., everyone was AAV5 negative.
Groups:
- BMN 270 (valoctocogene roxaparvovec): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg with prophylactic corticosteroids
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII, with Prophylactic Corticosteroids in Hemophilia A subjects
Period: Overall Study
Arm/Group | BMN 270 (valoctocogene roxaparvovec)
Started | 22
Continuing in the study | 22
Completed Week 52 visit | 22
Completed (Study is still ongoing.) | 0
Not Completed | 22

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population (N=22) - all participants who received BMN 270 infusion in 270-303 by the time of the data cutoff
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment, years
  years | 28.0 (7.4)
Age, Customized [Count of Participants; unit: Participants] — Age at enrollment: n(%)
  Participants
    18 to < 30 years | 13
    30 to < 50 years | 9
    >= 50 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Percentages were calculated using the total number of participants (N) in each analysis population as the denominator.
  Participants
    Female | 0
    Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — n(%)
  Participants
    Asian | 2
    Black or African-American | 2
    White | 18
Baseline annualized FVIII usage [Mean (Standard Deviation); unit: IU/kg/year] — The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25.
  IU/kg/year | 4342.74 (3184.01)
Baseline annualized number of FVIII infusions [Mean (Standard Deviation); unit: Infusions/year] — Annualized FVIII infusion rate (count/yr) = (sum(Number of FVIII replacement infusions during calculation period) /sum(follow-up days of the period))*365.25.
  Infusions/year | 149.13 (72.74)
Baseline ABR (treated bleeds) [Mean (Standard Deviation); unit: bleeds/year] — Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  bleeds/year | 5.61 (11.29)
Baseline ABR (treated bleeds) [Count of Participants; unit: Participants] — Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  Participants
    0 bleeds/year | 5
    >0 to 4 bleeds/year | 10
    >4 to 10 bleeds/year | 5
    >10 bleeds/year | 2
Baseline ABR (all bleeds) [Mean (Standard Deviation); unit: bleeds/year] — All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  bleeds/year | 8.20 (17.86)
Baseline ABR (all bleeds) [Count of Participants; unit: Participants] — All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  Annualized bleed rate (episodes/yr) = (sum (number of bleed episodes during calculation period))/(sum (follow-up days of the period)) *365.25
  Participants
    0 bleeds/year | 5
    >0 to 4 | 10
    >4 to 10 | 4
    >10 | 3
History of previous diseases [Count of Participants; unit: Participants] — Population: n(%)
  Participants
    Hepatitis B | 0
    Hepatitis C | 3
    HIV | 0
    No History of exposure to Hepatitis B/Hepatitis C/HIV | 19
Number of target joints [Count of Participants; unit: Participants] — n(%)
  Target joints are defined as joints with >= 3 spontaneous treated bleeds in the same joint location within any consecutive 6-month (180 days) period in the Baseline period.
  Participants
    0 | 16
    1 | 3
    2 | 2
    3 | 1
Adeno-associated virus Type 5 (AAV5) Total Antibody Titers and Positivity [Count of Participants; unit: Participants] — Percentages were calculated using the number of subjects with non-missing assessments (n) for each analysis population as the denominator.
  Participants
    Detected | 0
    Not detected | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FVIII Activity as Measured by Chromogenic Substrate Assay at Week 52.
Description: The change from baseline (assuming no treatment for severe hemophilia A) in FVIII activity, as measured by chromogenic substrate assay (CSA), at Week 52 (during Weeks 49 - 52) post-BMN 270 infusion.
  Each participant's FVIII activity level at Week 52 is defined as the median of the values obtained within the analysis window at Weeks 49-52. The baseline value will be imputed as 1 IU/dL, since there will be no washout of severe hemophilia A participants' usual FVIII prophylaxis (in order to avoid increasing the risk of bleeding) prior to BMN 270 infusion. Post-BMN 270 infusion values for FVIII activity will be excluded from analysis if obtained within 72 hours (or 3 calendar days if time is not available) since the last infusion of exogenous FVIII replacement therapy.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
Time Frame: Baseline to Week 52
Population: Modified intention-to-treat (mITT) population (N=21) - all participants who received BMN 270 infusion in 270-303 and were on adequate prophylactic hemophilia therapy for at least 12 months (adequate prophylaxis was defined as >= 52 doses of FVIII replacement therapy in 12 months if on FVIII prophylaxis) prior to BMN 270 infusion.
Measure: Mean (Standard Deviation); unit: IU /dL
Groups:
- BMN 270 (Valoctocogene roxaparvovec): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg with prophylactic corticosteroids
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A subjects
Arm/Group | BMN 270 (Valoctocogene roxaparvovec)
Number analyzed (Participants) | 21
IU /dL | 15.13 (22.38)
Statistical Analysis 1: Comparison: BMN 270 (Valoctocogene roxaparvovec); Test type: Superiority; p = 0.0057, t-test, 2 sided — P-value was based on two-sided t-test against 0

2. Secondary Outcome: Change From Baseline in Annualized Utilization of Exogenous FVIII Replacement Therapy in EEP
Description: The change from baseline (prior to BMN 270 infusion while receiving FVIII prophylaxis) in the annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy in the efficacy evaluation period ("Post-FVIII Prophylaxis period").
  The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for the analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to efficacy evaluation period (EEP)
Population: mITT population
Measure: Mean (Standard Deviation); unit: IU/kg/yr
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 21
IU/kg/yr | -4150.09 (3208.50)

3. Secondary Outcome: Change From Baseline in the Annualized Number of Bleeding Episodes Irrespective of Exogenous FVIII Replacement Treatment (Annualized Bleeding Rate, ABR for All Bleeds) in EEP
Description: All bleeds comprises both treated and non-treated bleeds. In this definition, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. All bleeds are any reported bleeding events regardless of the use of FVIII or other treatments.
  ABR for all bleeds= Number of bleeding episodes for all bleeds during the calculation period / total number of days during the calculation period * 365.25.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to efficacy evaluation period (EEP)
Population: mITT population
Measure: Mean (Standard Deviation); unit: bleeds/year
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 21
bleeds/year | -6.15 (17.24)

4. Secondary Outcome: Change From Baseline in the Annualized Number of Bleeding Episodes Requiring Exogenous FVIII Replacement Treatment (ABR for Treated Bleeds) in the EEP.
Description: ABR for treated bleeds=Number of bleeding episodes for treated bleeds during the calculation period/total number of days during the calculation period * 365.25
  Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis.
  EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or the end of FVIII prophylaxis plus the washout period (3 days for products of standard half-life or plasma-derived and 5 days for products of extended half-life), whichever is later, to last visit by the data cut-off for analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Time Frame: Baseline to EEP
Population: mITT population
Measure: Mean (Standard Deviation); unit: bleeds/year
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 21
bleeds/year | -3.78 (10.14)

5. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Total Score at Week 52
Description: The change from baseline(assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at wk52 post-BMN 270 infusion.The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life(HRQoL)questionnaire for adults consisting of 41 items covering 6 domains(Physical Functioning, Role Functioning,Worry,Consequences of Bleeding,Emotional Impact &Treatment Concerns). The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0(none of the time)to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-QoL-A domain(physical functioning, role functioning, worry, consequences of bleeding, emotional impact, treatment concern) scores range from 0 to 5 and the total score is derived by summing each domain score (range, 0 to 30). Domain and total scores are transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia related quality of life.
Time Frame: Baseline to Week 52
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 19
score on a scale | 6.70 (8.96)

6. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Physical Functioning Domain Score, at Week 52
Description: The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 52 post BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-Qol-A physical functioning domain score is an average of each item value within a domain.The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The physical functioning domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related physical functioning
Time Frame: Baseline to Week 52
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 19
score on a scale | 6.43 (8.51)

7. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Consequences of Bleeding Domain Score, at Week 52
Description: The change from baseline(assuming no treatment for severe hemophilia A)in Haemo-Qol-A score, at week 52 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life(HRQoL)questionnaire for adults consisting of 41 items covering 6 domains(Physical Functioning,Role Functioning,Worry,Consequences of Bleeding,Emotional Impact and Treatment Concerns). The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0(none of the time) to 5(all of the time). The recall period for the Haemo-Qol-A is one month (4-wks).
  The Haemo-Qol-A consequences of bleeding domain score is an average of each item value within a domain. The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The consequences of bleeding domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related consequences of bleeding.
Time Frame: Baseline to Week 52
Population: mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 19
score on a scale | 10.68 (16.33)

8. Secondary Outcome: Change From Baseline in Haemo-QoL-A Quality of Life: Role Functioning Domain Score, at Week 52
Description: The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 52 post BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time). The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-Qol-A role functioning domain score is an average of each item value within a domain. The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The role functioning domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related role functioning.
Time Frame: Baseline to Week 52
Population: mITT population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
Number analyzed (Participants) | 19
Score on a scale | 6.03 (10.29)

ADVERSE EVENTS:
Time Frame: Up to 112 weeks
Description: Intention-to-treat (ITT) population (N=22) - all participants who received BMN 270 infusion in 270-303 by the time of the data cutoff
Groups:
- BMN 270 (Valoctocogene Roxaparvovec): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg with prophylactic corticosteroids
  valoctocogene roxaparvovec: Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Hemophilia A
Arm/Group | BMN 270 (Valoctocogene Roxaparvovec)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 (Valoctocogene Roxaparvovec) (N=22)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 270 (Valoctocogene Roxaparvovec) (N=22)
Alanine aminotransferase increased (Investigations) | 20 (50)
COVID-19 (Infections and infestations) | 12 (12)
Acne (Skin and subcutaneous tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 7 (11)
Insomnia (Psychiatric disorders) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Influenza (Infections and infestations) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (9)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Influenza like illness (General disorders) | 3 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (9)
Agitation (Psychiatric disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Pregnancy of partner (Social circumstances) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Rash pustular (Infections and infestations) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT04323098/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04323098/SAP_001.pdf